CLINICAL TRIAL: NCT04399018
Title: Development and Prospective Validation of a Standardized Flow Cytometric Assay of Peripheral Blood Neutrophil Myeloperoxidase Expression for Ruling Out Myelodysplastic Syndromes.
Acronym: MPO-MDS-Develp
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC19.425; 2019-A03341-56 (Other: ID RCB)
Record Dates: First submitted 2020-05-18; First posted 2020-05-22 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Myelodysplastic Syndromes
Keywords: Diagnostic accuracy study; Flow cytometry analysis; Myeloperoxidase; Peripheral blood sample
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Diagnostic Test: Flow cytometry analysis of neutrophil myeloperoxidase expression — Flow cytometry analysis of neutrophil myeloperoxidase expression in peripheral blood samples will be performed within 24 h of MDS diagnostic evaluation and blinded to the reference standard. Peripheral blood samples will be collected in 5 ml (EDTA) anticoagulant plastic tubes and processed within 24 h maximum of collection.
  Blood sample will be stained according to the manufacturers' recommendations with a lyophilized cocktail ("LyotubeTM ready-to-use", BD Bioscience).
  At least 10,000 neutrophils will be acquired on a 3-laser, 8-color BD FACSCanto-II TM flow cytometer (BD Biosciences, San José, CA).
  Each marker will be expressed as median, geometric and arithmetic mean, regular and robust coefficient of variation.

SUMMARY:
Myelodysplastic syndromes (MDS) comprise a heterogeneous group of clonal bone marrow neoplasms that predominate in the elderly, with a median age at diagnosis of 70 years. The diagnosis of MDS relies on peripheral blood cytopenia and morphologic dysplasia for one or more hematopoietic cell lineage. Cytopenia is evidenced with hemogram while dysplasia requires bone marrow aspirate, which is an invasive procedure .

Considering the low prevalence of disease among subjects referred for suspected MDS, many patients are exposed to unnecessary bone marrow aspiration-related discomfort and harms. Therefore, an objective assay based on a peripheral blood sample that accurately discriminates MDS from other cytopenia etiologies is highly desirable.

We have previously developed and refined a flow cytometric analysis protocol for quantifying neutrophil MPO expression in peripheral blood at three university-affiliated hospitals (i.e., Clermont-Ferrand, Saint-Etienne, and Grenoble) (Raskovalova et al, Hematologica 2019). We found that the robust coefficient of variation (RCV, computed as the robust standard deviation divided by the median) within an individual subject was the best parameter in discriminating patients with versus without MDS.

Although promising, flow cytometric analysis of neutrophil MPO expression in peripheral blood is technically complex, time consuming, and not standardized. Hence, its performance requires specific expertise and the results show substantial variability. A single ready-to-use tube with lyophilized antibodies would have the potential to standardize the measurement of neutrophil MPO expression in peripheral blood across laboratories, with results available within 30-60 min in routine practice.

In this study, the investigators hypothesize that a standardized and semi-automatic flow cytometric assay of neutrophil MPO expression in peripheral blood could accurately rule out MDS and obviate the need for bone marrow aspiration and biopsy, with sensitivity and negative predictive value estimates approaching 100%.

In this observational diagnostic accuracy study, burden will be null for recruited patients. No specific intervention is assigned to participants. All diagnostic testing, procedures, and medication ordering are performed at the discretion of attending physicians. A test result will have no impact on patient management. .Compliance with current guidelines disseminated by the French Haute Autorité de Santé (HAS) will be advocated for the diagnostic work-up of patients with suspected MDS. No follow-up visits are planned in this cross-sectional study.

DETAILED DESCRIPTION:
The primary objective of MPO-MDS-develop study is to estimate the discriminative accuracy (i.e., area under the ROC curve along with 95% CI) of a standardized and semi-automatic flow cytometric assay of neutrophil MPO expression in peripheral blood for the diagnosis of MDS in adult patients.

The secondary objectives are to assess:

1. intra-laboratory reproducibility (intra- and inter-assay precision) for intra-individual RCV measurement of neutrophil MPO expression in peripheral blood;
2. specimen stability for intra-individual RCV measurement of neutrophil MPO expression in peripheral blood at different time points in comparison with H0 (stored at 4°C and at room temperature);
3. inter-laboratory reproducibility for intra-individual RCV measurement of neutrophil MPO expression in peripheral blood;
4. the negative predictive value for intra-individual RCV measurement of neutrophil MPO expression in peripheral blood (with a prespecified threshold of 30.0%) in ruling out MDS in consecutive adult patients.

The MPO-MDS-Develop project is a multicenter, cross-sectional, diagnostic accuracy study of an index test by comparison with a reference standard, in unselected consecutive patients.

Screening: All consecutive patients referred to the immuno-hematology lab at the study sites for suspicion of MDS will be screened for eligibility. A lab physician will review inclusion and exclusion criteria, using computerized medical and laboratory records.

Recruitment: Participants will be included in the study once all the screening activities have been conducted and only if the patient meets all inclusion and none exclusion criteria. The consent for flow cytometry analysis of peripheral blood sample and data collection through chart review will be sought under a regime of "non-opposition" (opt-out): after appropriate written information is delivered, cross-sectional data will be collected except in case of opposition from the patient. All patients included in the study will be assigned a unique patient identification number. This number will be used to identify the patient throughout the study.

Index test: Flow cytometry analysis of neutrophil myeloperoxidase expression in peripheral blood will be performed using a single ready-to-use tube with lyophilized antibodies developed in partnership with Becton Dickinson France SAS and blinded to the reference standard.

Reference standard: The diagnosis of MDS will be established according to the World Health Organization (WHO) classification, based on clinical data, peripheral blood cytopenia, cytomorphology of peripheral blood and bone marrow aspirate, and cytogenetic analysis. The criteria for MDS diagnosis are 1) the presence of ≥10% dysplastic cells in any hematopoietic lineage, 2) the exclusion of acute myeloid leukemia (defined by the presence of ≥20% peripheral blood or bone marrow blasts), and 3) the exclusion of reactive etiologies of dysplasia. Cytopenia is defined by hemoglobin concentration <10 g/dL, platelet count <100x109/L, and/or absolute neutrophil count <1.8 x109/L. Yet a diagnosis of MDS could be made with milder levels of cytopenia. Idiopathic cytopenia of uncertain significance (ICUS) is defined by unexplained mild persistent cytopenia for at least 6 months and the failure to establish the diagnosis to MDS according to published guidelines. Consistent with WHO classification, MDS subcategorization will rely on the degree of dysplasia (unilineage versus multilineage), blast percentages, presence of ring sideroblasts, and cytogenetic analysis (del(5q)). The criteria for CMML diagnosis are 1) the presence of persistent peripheral blood monocytosis ≥1 x109/L, and 2) monocyte accounting for more than 10% of the white blood cell differential count. Evaluation of bone marrow cytomorphology will be performed prospectively by experienced hematopathologists who are blinded to the index test results.

Patients with confirmed suspicion of MDS: Participants for whom the diagnosis of MDS (or CMML) is confirmed by the reference standard will be categorized as patients with confirmed suspicion of MDS.

Patients with unconfirmed suspicion of MDS: Participants for whom the diagnosis of MDS (or CMML) is ruled out by the reference standard will be categorized as patients with unconfirmed suspicion of MDS. This latter subgroup will include patients with ICUS, as defined in accordance with published guidelines.

Follow-up: No follow-up visit is planned in this cross-sectional diagnostic accuracy study.

ELIGIBILITY:
Inclusion Criteria:

* Age at enrollment ≥18 years
* Clinical suspicion of MDS
* Indication for bone marrow examination
* ≥1 peripheral blood cytopenia defined by hemoglobin concentration <12 g/dL for female and <13g/dL for male patients, platelet count <150 x109/L, absolute neutrophil count <1.8 x109/L
* Inpatient and outpatient care patients

Exclusion Criteria:

* Refusal to participate
* History of or active documented MDS
* Enrollment in intensive or critical care unit
* Incarcerated or individuals protected by French regulation (Article L1121.5 and following, Code de la Santé Publique)
* Not affiliated with social security system
* Previous enrollment in the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants are unselected consecutive adults referred for suspected MDS. Suspicion of MDS is based on medical history and peripheral blood cytopenia. To be eligible, patients will be required to meet all five inclusion criteria and none of the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Reference diagnosis of MDS or CMML established by bone marrow examination | Baseline
  The primary outcome is the reference diagnosis of MDS or CMML established by bone marrow examination (with Perls staining) by two independent experienced hematopathologists blinded to the index test results. Disagreements will be solved by a third hematopathologist. Bone marrow aspirate will be repeated within 4 to 6 months for patients with idiopathic cytopenia of uncertain significance (ICUS) or non-conclusive bone marrow examination.

SECONDARY OUTCOMES:
Intra-laboratory coefficient of variation for intra-individual RCV, computed as the standard deviation multiplied by 100 and divided by the mean (intra- and inter-assay precision) | Baseline
Relative change from baseline, expressed in percentages for intra-individual RCV | Baseline
Inter-laboratory coefficient of variation for intra-individual RCV | Baseline
Negative predictive value point estimates (along with 95% confidence interval) of neutrophil myeloperoxidase expression in peripheral blood for the diagnosis of MDS or CMML | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Raskovalova, MD, Study Chair — Centre Hospitalier Universitaire Grenoble Alpes; Richard Veyrat-Masson, MD, Principal Investigator — Centre Hospitalier Universitaire Clermont Ferrand; Carmen Aanei, MD, Principal Investigator — Centre Hospitalier Universitaire Saint-Étienne
Locations (1):
- Chu Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: Yes
The principal investigators will respond directly to data requests by providing a de-identified data set. Individual participant data that underlie the results reported in the published articles (i.e., main text, tables, figures, and appendices) will be supplied.
Supporting Information: Study Protocol, SAP
Time Frame: No later than 3 years after final acceptance of the primary study paper.
Access Criteria: De-identified data will be available for individual participant data meta-analysis purpose.
  Researchers should submit a methodologically sound proposal that complies with the Preferred Reporting Items for Systematic Review and Meta-Analysis Protocols (PRISMA-P) 2015 statement. Proposals should be directed to TRaskovalova@chu-grenoble.fr. Data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Planta C, Scheffen L, Jacob MC, Szymanski G, Chevalier S, Tondeur S, Bulabois B, Meunier M, Lefebvre C, Gonnet N, Garban F, Molina L, Paradis C, Seigneurin A, Chiriac R, Merle R, Labarere J, Park S, Raskovalova T. Flow cytometric lyophilised reagent tube assay for peripheral blood neutrophil myeloperoxidase expression to rule out myelodysplastic neoplasms at a university hospital: a diagnostic accuracy study. BMJ Open. 2025 Aug 22;15(8):e095640. doi: 10.1136/bmjopen-2024-095640. PMID 40846335
- [Derived] Raskovalova T, Scheffen L, Jacob MC, Chevalier S, Tondeur S, Bulabois B, Meunier M, Szymanski G, Lefebvre C, Planta C, Dumestre-Perard C, Gonnet N, Garban F, Merle R, Park S, Labarere J. Flow cytometry lyophilised-reagent tube for quantifying peripheral blood neutrophil myeloperoxidase expression in myelodysplastic syndromes (MPO-MDS-Develop): protocol for a diagnostic accuracy study. BMJ Open. 2022 Oct 7;12(10):e065850. doi: 10.1136/bmjopen-2022-065850. PMID 36207039